CLINICAL TRIAL: NCT04693845
Title: Aftercare Focus Study (AFS): A Clinical Trial to Reduce Short-Term Suicide Risk After Hospitalization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Catholic University of America (Other); American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Kate Comtois, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00010396
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Distress, Psychological; Quality of Life
Keywords: Suicidal Ideation; Suicide, Attempted; Distress, Psychological; Psychotherapy
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Community Mental Health Center Next Day Appointment clinic
  Interventions: Behavioral: Treatment as Usual
- Experimental (Experimental): Collaborative Assessment and Management of Suicidality (CAMS)
  Interventions: Behavioral: Collaborative Assessment and Management of Suicidality

INTERVENTIONS:
Behavioral: Collaborative Assessment and Management of Suicidality — CAMS is a suicide-focused intervention that stabilizes the suicidal patient and identifies, targets, and treats patient-defined "suicidal drivers"-the problems (e.g., trauma, financial issues, relationship loss) that compel a patient to consider suicide. CAMS is theoretically agnostic, patient-centered, and can be used across different suicidal populations and clinical settings.
  Arms: Experimental
Behavioral: Treatment as Usual — Treatment as Usual was based on the staff, policies, and procedures of the community mental health center Next Day Appointment clinic (CMHC) affiliated with our university. Research therapists and the research psychiatrist were hired from the CMHC staff who followed standard CMHC policies and procedures.
  Arms: Treatment as Usual

SUMMARY:
Increasingly, the period after hospital admission is acknowledged as one of extremely high risk for suicidal patients. While it might be hoped that hospitalization would address and resolve suicide risk, a review of international studies shows the risk of suicide is up to 200 times higher among individuals recently discharged from hospitals vs. the general population. In response, some health care systems use an "urgent care" or "next-day appointment" (NDA) clinics for follow-up. NDAs serve as short-term crisis intervention at a specific appointment time and location so patients do not "fall through the cracks" in the care transition. Collaborative Assessment and Management of Suicidality (CAMS) is a potentially effective intervention to reduce short term suicidal risk in this transition from inpatient to outpatient treatment. To this end, this study has the following study aims: (1) Evaluate whether CAMS for suicidal NDA patients results in less suicidal behavior than TAU, (2) Evaluate whether CAMS for suicidal NDA patients results in less suicidal ideation and intent as well as improved mental health markers than TAU, and (3) Evaluate whether CAMS for suicidal NDA patients is more satisfactory to patients than TAU.

DETAILED DESCRIPTION:
Increasingly, the period after hospital admission is acknowledged as one of extremely high risk for suicidal patients. While it might be hoped that hospitalization would address and resolve suicide risk, a review of international studies shows the risk of suicide is up to 200 times higher among individuals recently discharged from hospitals vs. the general population. In response, some health care systems use an "urgent care" or "next-day appointment" (NDA) clinics for follow-up. NDAs serve as short-term crisis intervention at a specific appointment time and location so patients do not "fall through the cracks" in the care transition. Collaborative Assessment and Management of Suicidality (CAMS) is a promising outpatient treatment framework that merits rigorous study as a potentially effective intervention to reduce short term suicidal risk in the transition from inpatient to outpatient treatment. Pilot data suggest that CAMS decreases suicidal ideation and psychological distress while increasing hope, patient satisfaction, and retention more than NDA treatment as usual (TAU). CAMS in the NDA clinic has the potential to fill three key targets highlighted in the 2012 National Strategy for Suicide Prevention: (1) prevent suicidal behavior, (2) increase clinician confidence and willingness to see suicidal patients, and (3) are sufficiently feasible, trainable, adaptable, and flexible to scale up across health systems. To this end, this study has the following study aims: (1) Evaluate whether CAMS for suicidal NDA patients results in less suicidal behavior than TAU, (2) Evaluate whether CAMS for suicidal NDA patients results in less suicidal ideation and intent as well as improved mental health markers than TAU, and (3) Evaluate whether CAMS for suicidal NDA patients is more satisfactory to patients than TAU.

ELIGIBILITY:
Inclusion Criteria:

1. inpatient or emergency service admission for suicidality or suicide attempt
2. lifetime suicide attempt
3. referring clinician determined that the patient did not have appropriate outpatient mental health appointment in the next two weeks (other than an NDA)
4. an NDA is an appropriate disposition plan
5. consented to all study procedures.

Exclusion Criteria:

1. under age 18
2. insufficient English to understand the study procedures and provide informed consent
3. too psychotic or manic, aggressive, or cognitively impaired such that outpatient therapy was not indicated
4. patient not stable enough to be discharged home for a minimum of 24 hours prior to study treatment
5. court-ordered to outpatient treatment
6. patient lived an impractical distance away

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Suicidal behavior | Twelve months
  Suicidal behavior will be a count of a suicide + all suicide attempts + all acute hospitalizations to prevent suicide. Suicide will be determined by death records; Suicide attempts measured with the Suicide Attempt Self-Injury Count; Hospitalizations measured with the Treatment History Interview-Short Form
Suicidal ideation | Twelve months
  Beck Scale for Suicidal Ideation (BSS) (19 item scale scored 0-2 so scores range from 0-38 with higher scores indicating worse ideation)
Suicidal intent | Twelve months
  Beck Suicide Intent Scale (SIS) (17 item scale scored 0-2 so scores range from 0-34 with higher scores indicating stronger suicide intent)
Psychological Distress | Twelve months
  Outcome Questionnaire-45.2 (45 item scale scored 0-4 with three subscales (symptom distress, interpersonal problems, and social role functioning) and a total score ranging from 0-180 with higher scores indicating worse outcomes)
Quality of life and overall functioning | Twelve months
  EQ-5D (5 items scored using an algorithm to create an index value anchored at 1=full health and 0=dead)(Note the measure of this construct was changed from proposed Lehman Quality of Life Interview prior to study recruitment to reduce subject burden)
Treatment Satisfaction | Through the end of study treatment, an average of 3 months
  Client Satisfaction Questionnaire (8 item scale scored 1-4 resulting in a score ranging from 1-32 with higher indicating greater satisfaction with treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Comtois, PhD, MPH, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No